CLINICAL TRIAL: NCT07020156
Title: A First in Human Phase 1 Trial of OX118 in Healthy Volunteers
Brief Title: A First-in-Human Phase I Trial of OX118 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oxion Biologics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SAPIOX
Record Dates: First submitted 2025-04-02; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Immune System

STUDY DESIGN:
Intervention Model Description: Cohort 1: 0.1 mg/kg OX118 or placebo (3:1) Cohort 2: 0.3 mg/kg OX118 or placebo (3:1) Cohort 3: 1 mg/kg OX118 or placebo (6:2) Cohort 4: 3mg/kg OX118 or placebo (6:2) Cohort 5: 10mg/kg OX118 or placebo (6:2)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental or placebo 0,1mg/kg (3:1) (Experimental): IMP: OX118 Number of participants: 4 Route of administration: intravenous infusion
  Interventions: Drug: OX118 or placebo
- Experimental or placebo 0,3mg/kg (3:1) (Experimental): IMP: OX118 Number of participants: 4 Route of administration: intravenous infusion
  Interventions: Drug: OX118 or placebo
- Experimental or placebo 1mg/kg (6:2) (Experimental): IMP:OX118 Number of participants: 8 Route of administration: intravenous infusion
  Interventions: Drug: OX118 or placebo
- Experimental or placebo 3mg/kg (6:2) (Experimental): IMP:OX118 Number of participants: 8 Route of administration: intravenous infusion
  Interventions: Drug: OX118 or placebo
- Experimental or placebo 10mg/kg (6:2) (Experimental): IMP:OX118 Number of participants: 8 Route of administration: intravenous infusion
  Interventions: Drug: OX118 or placebo

INTERVENTIONS:
Drug: OX118 or placebo — OX118 is a human monoclonal antibody targeting OX40 ligand (OX40L).

SUMMARY:
This is a first-in-human, phase 1 study of OX118 in healthy volunteers, designed to investigate the safety and tolerability of OX118, as well as its pharmacokinetics (the drug's concentration in the blood and excretion from the body).

The study will include a total of 32 participants: healthy men and women aged 18-60 years with a body mass index (BMI) between ≥18.5 and ≤30.0.The study is divided into five cohorts where OX118 will be given as a single dose intravenously (into the blood).

The study consists of 7 clinic visits taking place over a period of approximately 77 days (including a 28-day screening period). During the study, subjects will be given the study drug (OX118) or placebo. Both the study drug and the placebo will be given as a single dose as an intravenous (directly into the blood) infusion. A pre-arranged schedule will determine whether subjects will receive the study drug or the placebo.

DETAILED DESCRIPTION:
Participants will recieve either OX118 or placebo.

* Cohort 1: 0.1 mg/kg OX118 or placebo (3:1)
* Cohort 2: 0.3 mg/kg OX118 or placebo (3:1)
* Cohort 3: 1 mg/kg OX118 or placebo (6:2)
* Cohort 4: 3mg/kg OX118 or placebo (6:2)
* Cohort 5: 10mg/kg OX118 or placebo (6:2)

Each participant is expected to take part in the trial for approximately 91 days, including an up to 28-day screening period. Participants will come for 7 visits to the research clinic for screening, treatment, and follow-up (visit 2 including two nights at the clinic).

Sentinel dosing will apply to the first 2 participants in each cohort, except for the first cohort where the first 2 participants will be dosed separately in order to maintain the blind. All Participants will remain in the trial site for 24 hours after IMP administration and will be closely monitored by medical staff. Visits at the site may be prolonged in the event that the Investigator finds it medically warranted for safety reasons.

Safety assessments

* AEs
* IRRs
* Vital signs (supine blood pressure [BP]), pulse, body temperature)
* 12-lead ECG
* Safety laboratory assessments (haematology, clinical chemistry and coagulation)
* Physical examinations
* Concomitant mediations

Once safety and tolerability data up until and including 7 days in the previous cohort have been collected and all participants have been dosed, all treated participants must have been reviewed by the internal safety review committee (iSRC) before a new cohort may be initiated. Based on emerging safety and tolerability, the amount of required data to be reviewed after each completed cohort may be adjusted.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the trial.
2. Healthy male or female participant aged 18 to 60 years, inclusive.
3. Weighs ≥ 50 and ≤ 100 kg and has a body mass index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2 at the time of the screening visit.
4. Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values at the time of the screening visit, as judged by the Investigator.

   (Discussion is encouraged between the Investigator and the Sponsor medical representative regarding the clinical relevance of any abnormal laboratory value during the pre-dose period.)
5. Women of childbearing potential (WOCBP) must practice abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the participant) or must agree to use a highly effective method of contraception with a failure rate of <1 % to prevent pregnancy from at least 2 weeks prior to the administration of IMP to 3.5 months (15 weeks) after the last administration of IMP. In addition, any male partner of a female participant must, unless he has undergone vasectomy, agree to use a condom from the administration of IMP until 3.5 months (15 weeks) after the last administration of IMP.

The following are considered highly effective methods of contraception:

* combined (oestrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal),
* progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable),
* intra-uterine device [IUD]or intra-uterine hormone-releasing system [IUS]). WOCBP must refrain from donating eggs from the first IMP administration until 6 months after the last IMP administration. WOCBP with an exclusive male partner who has undergone vasectomy may choose not to use contraceptives.

Women of non-childbearing potential are pre-menopausal females who have undergone any of the following surgical procedures; hysterectomy, bilateral salpingectomy or bilateral oophorectomy, or who are post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] >25 IU/L is confirmatory).

Male participants must be willing to use a condom or be vasectomised or practice sexual abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the participant) to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the first administration of IMP until 6 months after the last administration of IMP. Any female partner of a non-vasectomised male participant who is of childbearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above) from at least 2 weeks prior to the first administration of IMP to 3.5 months (15 weeks) after the last administration of IMP

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial or influence the results or the participant's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the administration of IMP.
3. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the trial.
5. Participants who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
6. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis C antibodies and/or human immunodeficiency virus (HIV).
7. After 10 minutes supine rest at the screening visit, any vital signs values outside the following ranges:

   * Systolic BP: <90 or ≥140 mmHg, or
   * Diastolic BP <50 or ≥90 mmHg, or
   * Pulse <40 or ≥90 bpm
8. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the screening visit, as judged by the Investigator.
9. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to OX118.
10. Regular use of any prescribed or non-prescribed medications, including antacids, analgesics, herbal remedies, vitamins and minerals, within 2 weeks prior to the administration of IMP, except occasional intake of paracetamol (maximum 2000 mg/day and not exceeding 3000 mg/week), as well as nasal decongestants without cortisone, antihistamine or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
11. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1. Participants who consented and screened but were not dosed in previous Phase I trials are not to be excluded.
12. Current smokers or users of nicotine products (e.g., smoking, snuffing, chewing tobacco) corresponding to ≥ 5 cigarettes per day.
13. Positive screening result for drugs of abuse or alcohol at the screening visit or on admission to the trial site prior to the administration of the IMP. (Positive results that are expected given the participant's medical history and prescribed medications can be disregarded as judged by the Investigator.)
14. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
15. Presence or history of drug abuse, as judged by the Investigator.
16. History of, or current use of anabolic steroids, as judged by the Investigator.
17. Excessive caffeine consumption defined by a daily intake of > 5 cups (1 cup = approximately 240 mL) of caffeine-containing beverages, as judged by the Investigator.
18. Plasma donation within 1 month of screening or blood donation (or corresponding blood loss) during the last 3 months prior to screening.
19. The Investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] [Time Frame: Day 1 to Day 63] | Day 1 to Day 63
  To evaluate the safety and tolerability of OX118 following single IV SAD administration in healthy male and female volunteers
Number of Participants with Abnormal Vital Signs | Day 1 to Day 63
Number of Participants With Abnormal Laboratory Values | Day 1 to Day 63
Number of Participants with Abnormal Electrocardiograms (ECGs) | Day 1 to Day 63
Number of Participants with Abnormal Physical Examination Findings | Day 1 to Day 63

SECONDARY OUTCOMES:
AUC | Day 1 to Day 63
  Area under the plasma concentration vs. time curve (AUC).
Cmax | Day 1 to Day 63
  Maximum plasma concentration (Cmax).
Tmax | Day 1 to Day 63
  Time to Cmax (Tmax).
Cl | Day 1 to Day 63
  Clearance.
Vz | Day 1 to Day 63
  Apparent volume of distribution associated with terminal slope
Vss | Day 1 to Day 63
  An estimation of the apparent volume of distribution at steady state
Tlast and AUCextr | Day 1 to Day 63
  Percentage extrapolated from time of occurrence of the last observed plasma concentration (Tlast) to infinity (AUCextr).
Evaluate immunogenicity of IMP after IV administration. | Day 1 to Day 63
  To evaluate the immunogenicity of OX118 following IV SAD administration in healthy male and female volunteers. Incidence of anti-drug antibodies (ADAs) directed against OX118 as measured by titers of anti-OX118 in serum.
Immune phenotype | Day 1 to Day 63
  Immune system composition in peripheral blood (i.e., immune phenotyping [IPT]).

CONTACTS AND LOCATIONS:
Locations (1):
- CTC, Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided